CLINICAL TRIAL: NCT00911690
Title: Establishment of a Bank of Biospecimens for the Evaluation of New Methods Facilitating Early Diagnosis and the Monitoring of Progression and Therapy of Patients With Age-related Cognitive Disorders.
Brief Title: Establishment of a Bank of Biospecimens for Future Research on Age-related Cognitive Disorders
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Khaled Imam, Director, Division of Geriatric Medicine, Corewell Health East
Other Study IDs: 2008-065
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Dementia; Alzheimers Disease
Keywords: Dementia; Alzheimers Disease; Cognitive Disorders; Tissue Banking
MeSH Terms: conditions — Dementia; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, human platelet, urine (clarified), urine sediment, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cognitively Impaired: Patients in this cohort with be diagnosed with mild to moderate cognitive impairment, Alzheimers disease, Dementia, or any other form of cognitive impairment.
- Non-cognitively impaired: Patients in this cohort will be normal healthy adults over the age of 60 years that have no cognitive impairment.

SUMMARY:
This study is collecting tissue specimens (blood, urine and saliva) from up to 1000 patients, with and without cognitive disorders, to store in the Bio Bank for future research. The specimens could be used in future research projects that could help improve the accuracy of diagnosis of a disease, predict who might develop a disease, help monitor the disease, or improve the understanding of the disease. Patients are only being recruited from Beaumont Hospitals Geriatric Clinic.

DETAILED DESCRIPTION:
Up to 1000 patients, with or without diagnosed cognitive disorders, are asked to participate by providing the investigators with blood, urine and saliva specimens to be stored in a Bio Bank for future research. Patients will be asked to participate on a yearly basis for up to 5 to 10 years by providing the investigators with the above-mentioned specimens, and also having a physical exam and having some cognitive testing performed at the initial visit and yearly visits.

Examples of the types of research are: new methods for improving the diagnosis and treatment of age-related cognitive disorders, new areas of biology, new areas of biotechnology, and possibly genetic research. If you do not want your specimens used for any specific type of research, you may specify that on the consent form.

ELIGIBILITY:
Inclusion Criteria:

1. At least 60 years of age.
2. Willing and able to complete all specimen donations and neuropsychological examinations.
3. Individuals identified as having some form of cognitive impairment require a study partner with 1-2 times per week contact (can be in person and/or telephone), who will accompany them to study visits(s).

Exclusion Criteria:

1. Presence of significant sensory deficits (e.g., visual or hearing), motor deficits (e.g., paralysis), or medical conditions that would preclude the completion of the neuropsychological or other study instruments.
2. DMS-IV diagnosis of substance abuse disorder.
3. Presence of a major medical or terminal illness that may affect the participation of the patient in the study.
4. Known active malignancy, or history of malignancy within the last 5 years (other than basal cell carcinoma), severe organ failure, metabolic or hematologic disorders, or post-encephalitic syndrome.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be obtained from individuals seen by the physicians affiliated with the Division of Geriatric Medicine at Beaumont Hospital in the Geriatric Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2009-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Tissue bank of biological specimens | 5-10 years
  To establish a tissue bank of blood, urine and saliva from cognitively normal and cognitively impaired individuals 60 years or older to be used for the purpose of conducting research addressing: etiology, mechanism, diagnosis, and treatment of age-related cognitive disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Imam, M.D., Principal Investigator — Beaumont Hospitals
Locations (1):
- Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
If IPD are shared, it will be results of genomic and proteomic testing. As this testing was done throughout the study and is ongoing, some results are already available. Anyone interested would contact the principal investigator.